CLINICAL TRIAL: NCT06202443
Title: Improving Surgical Outcomes With Early Physical Therapy After Anterior Cervical Discectomy and Fusion
Brief Title: Function After Anterior Cervical Discectomy and Fusion Surgery: Timing of Physical Therapy (FAST-PT)
Acronym: FAST-PT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristin Archer, Professor and Vice Chair, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 231031
Record Dates: First submitted 2023-12-28; First posted 2024-01-11 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cervical Spine Degeneration; ACDF Surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Physical Therapy (PT) (Experimental): PT will be delivered two times a week for 8 weeks by a licensed physical therapist. Participants will start PT approximately 2 weeks after hospital discharge
  Interventions: Other: Early PT
- Delayed Physical Therapy (PT) (Active Comparator): PT will be delivered two times a week for 8 weeks by a licensed physical therapist. Participants will start PT approximately 3 months after hospital discharge.
  Interventions: Other: Delayed PT

INTERVENTIONS:
Other: Early PT — Physical therapy delivered within the first three months after surgery.
  Arms: Early Physical Therapy (PT)
Other: Delayed PT — Physical therapy delivered greater than 3 months after surgery.
  Arms: Delayed Physical Therapy (PT)

SUMMARY:
The goal of this two-group randomized clinical trial is to examine the effects of early postoperative PT compared to delayed postoperative PT for improving outcomes after hospital discharge for ACDF surgery.

The main question this clinical trial aims to answer are:

* Whether early PT participants will demonstrate greater improvements in outcomes compared to delayed PT participants.
* Whether improvements in handgrip strength, cervical endurance, and cervical range of motion will be associated with improvements in outcomes.

Participants will be randomized to one of two groups (early PT or delayed PT) and outcomes compared across groups.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial of early PT (within 3 months after surgery) versus delayed PT (greater than 3 months after surgery) in adults following ACDF surgery for degenerative conditions. The central hypothesis is that an early PT program will be effective in improving disability, pain, physical function, opioid use and return to work/duty. 76 participants will be enrolled and randomized (38 patients per randomized group), with 64 (85%) expected to be retained in the trial at the 12-month follow-up. Eligible patients undergoing ACDF surgery for a degenerative condition will be randomized to one of two groups (early PT or delayed PT). Patients will be enrolled prior to surgery, asked to complete a preoperative questionnaire prior to surgery and then randomized. Patients randomized to one of the PT groups will have their first PT visit scheduled for them by study staff prior to surgery. This visit will occur at approximately 2 weeks after hospital discharge for the early PT group and approximately 3 months after hospital discharge for the delayed PT group. All randomized patients will be asked to participate in follow-up visits approximately 3-, 6- and 12-months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Surgical treatment of a cervical degenerative condition using a 1- or 2-level ACDF procedure;
* English speaking due to feasibility of employing study personnel to deliver and assess the study intervention; and
* Age 18-75 years of age (individuals older than 75 are more likely to experience respiratory and nervous system complications and death following ACDF)

Exclusion Criteria:

* Surgery secondary to trauma, fracture, tumor, infection, or spinal deformity;
* Undergoing cervical corpectomy;
* Prior history of cervical spine surgery in last 5 years;
* Diagnosis or presence of osteoporosis;
* Diagnosis or presence of severe psychiatric disorder such as schizophrenia or bipolar disorder;
* Documented history of alcohol and/or drug abuse;
* Currently involved in litigation due to injury;
* Currently undergoing treatment for cancer;
* Patients not able to return for follow-up visits due to time and travel limitation or other reasons; and
* Unable to provide a stable telephone or physical address

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Disability | 6 and 12 months after hospital discharge
  Neck Disability Index, 0-100 with higher scores indicating increased disability

SECONDARY OUTCOMES:
Pain Intensity | 6 and 12 months after hospital discharge
  Numeric Rating Scale, 0-10 with higher scores indicating increased pain intensity
Pain Interference | 6 and 12 months after hospital discharge
  PROMIS, 0-100 with higher scores indicating increased pain interference
Physical Function | 6 and 12 months after hospital discharge
  PROMIS, 0-100 with higher scores indicating better physical function
Opioid Utilization | 6 and 12 months after hospital discharge
  MMEs
Return to work | 6 and 12 months after hospital discharge
  Work Productivity and Activity Impairment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Archer, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (4):
- United States (4):
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Booke Army Medical Center, Fort Sam Houston, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coronado RA, Devin CJ, Pennings JS, Aaronson OS, Haug CM, Van Hoy EE, Vanston SW, Archer KR. Safety and feasibility of an early telephone-supported home exercise program after anterior cervical discectomy and fusion: a case series. Physiother Theory Pract. 2021 Oct;37(10):1096-1108. doi: 10.1080/09593985.2019.1683921. Epub 2019 Oct 30. PMID 31663795
- [Background] Coronado RA, Devin CJ, Pennings JS, Vanston SW, Fenster DE, Hills JM, Aaronson OS, Schwarz JP, Stephens BF, Archer KR. Early Self-directed Home Exercise Program After Anterior Cervical Discectomy and Fusion: A Pilot Study. Spine (Phila Pa 1976). 2020 Feb 15;45(4):217-225. doi: 10.1097/BRS.0000000000003239. PMID 31490861